CLINICAL TRIAL: NCT05850546
Title: Efficacy and Safety of Single-dose Rituximab Biosimilar in the Initial Episode of Paediatric Steroid-sensitive Nephrotic Syndrome: A Multicenter, Open-Label, Noninferiority, Randomized Controlled Trial
Brief Title: Rituximab in the First Episode of Paediatric Nephrotic Syndrome
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Shen Kang Hospital Development Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Children's Medical Center (Other); Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTXFIRPedINS2
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Steroid-Sensitive Nephrotic Syndrome
Keywords: Rituximab; Children; Relapse
MeSH Terms: conditions — Nephrotic Syndrome; Recurrence | interventions — Rituximab; Adrenal Cortex Hormones; Prednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): Rituximab (375 mg/m2) will be given as a single intravenous infusion after remission. The prednisolone at a dose of 2 mg/kg per day (maximum 60 mg in single or divided doses) for 6 weeks, followed by 1.5 mg/kg (maximum 40 mg) as a single morning dose on alternate days for the next 6 weeks; therapy is then discontinued.
  Interventions: Drug: Rituximab; Drug: Corticosteroid
- Routine Therapy (Other): The prednisolone at a dose of 2 mg/kg per day (maximum 60 mg in single or divided doses) for 6 weeks, followed by 1.5 mg/kg (maximum 40 mg) as a single morning dose on alternate days for the next 6 weeks; therapy is then discontinued.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 added to guideline-recommended corticosteroid therapy
  Other Names: rituximab biosimilar (HANLIKANG®, Shanghai Henlius Biotech, Inc. China)
  Arms: Rituximab
Drug: Corticosteroid — guideline-recommended corticosteroid therapy
  Other Names: prednisolone/prednisone

SUMMARY:
The study will be a randomized, open-label trial in children with the initial episode of SSNS and whose state of complete remission after received standard prednisolone, to determine whether rituximab (a single intravenous infusion of 375 mg/m2) would be noninferior to corticosteroid alone in maintaining complete disease remission during 12-month of follow-up.

DETAILED DESCRIPTION:
The 12-month relapse-free survival rate is less than 30% in steroid-sensitive nephrotic syndrome (SSNS) children after the standard corticosteroid therapy, with approximately half becoming frequent relapsers or steroid dependent and necessitating the need for alternative immunosuppressive agents. The first relapse of SSNS most occurs within 6-12 months of onset, and contemporary cohorts suggest up to 16-42% of children with SSNS continue to have relapses in adulthood. Rituximab and rituximab biosimilar appear effective in reducing the relapse in children with frequent relapse or steroid dependent nephrotic syndrome. Accordingly, we hypothesize in paediatric SSNS, rituximab added to guideline-recommended corticosteroid therapy is noninferior to corticosteroid alone for maintaining remission for the first year of onset, expected to improve long-term outcomes.

An open-label, single-arm, multicentre trial was performed at eight centers in China with a 12-month follow-up (NCT04783675). The study found that in children with the initial episode of SSNS, rituximab appears to be an effective and safe treatment for maintaining disease remission.

The goal of this prospective study is to determine whether rituximab (a single intravenous infusion of 375 mg/m2) would be noninferior to corticosteroid alone in maintaining complete disease remission during 12-month of follow-up. The study will be a randomized, open-label, parallel group, in a 1:1 ratio, active controlled, multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 1 and 18 years with Steroid-Sensitive Nephrotic Syndrome (nephrotic-range proteinuria and either hypoalbuminemia or edema when albumin level is not available)
2. Estimated glomerular filtration rate (eGFR) ≥90 ml/min per 1.73 m2 at study entry
3. Remission at study entry
4. the cluster of differentiation antigen 20 (CD20) positive cells in peripheral blood ≥1% total lymphocytes
5. No immunosuppressive agents have been used within 3 months of enrolment, except for the use of corticosteroid to treat nephrotic syndrome
6. Provision of consent by a legal representative using a document approved by the institutional review board after receiving an adequate explanation of this clinical trial. For children ages 8-18, written assent is required using age-appropriate and background-appropriate documents

Exclusion Criteria:

1. Diagnosis of secondary NS
2. Patients showing one of the following abnormal clinical laboratories
3. values: leukopenia (white blood cell count ≤3.0*109/L); moderate and severe anemia (hemoglobin <9.0g/dL); thrombocytopenia (platelet count <100*1012/ L); positivity of autoimmunity tests (ANA, Anti DNA antibody, ANCA) or reduced C3 levels; Alanine aminotransferase or aspartate aminotransferase > 2.5× upper limit of normal value
4. Presence of severe or chronic infections within 6 months before assignment: tuberculosis or in whom tuberculosis is suspected; Epstein-Barr virus or cytomegalovirus; hepatitis B or hepatitis C or hepatitis B virus carrier, human immunodeficiency virus or other active viral infections
5. Live vaccination within last month
6. Patients with poorly controlled hypertension
7. Patients with severe brain, heart, liver, and other important organs, as well as blood and endocrine system diseases
8. Presence or history of autoimmune diseases, primary immunodeficiency, or tumor
9. Patients with a known allergy to Rituximab and its excipients
10. Assessed to be unfit for participation by the investigators (patients highly likely to be lost to follow-up or provide inaccurate data, for example, patients with alcohol or other substance misuse disorders, and patients with psychological disorders)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
1-year relapse-free survival rate | 1-year after randomization
  The rate of no relapse within 1 year. Relapse definition: recurrence of nephrotic-range proteinuria, urine protein/creatinine ratio ≥2 mg/mg or dipstick ≥3+ on 3 consecutive days in the first morning samples.

SECONDARY OUTCOMES:
Time to relapse (days) | 1-year after randomization
  Number of days from randomization to occurrence of first relapse. Relapse definition: recurrence of nephrotic-range proteinuria, urine protein/creatinine ratio ≥2 mg/mg or dipstick ≥3+ on 3 consecutive days in the first morning samples.
Peripheral blood T cell subsets | At basline, 1,3,6,9,12 months after randomization
  It is a repeat measured variable. Using fluorescence-activated cell sorting, peripheral blood T cells subsets will be studied as percentages and absolute counts.
Peripheral blood B cell subsets | At basline, 1,3,6,9,12 months after randomization
  It is a repeat measured variable. Using fluorescence-activated cell sorting, peripheral blood B cells subsets will be studied as percentages and absolute counts.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1-year after randomization
  It is a binary variable (1/0). The variable would be setted as "1" if any adverse events occurs including infusion- related reactions, infection (upper respiratory tract infection, hepatitis B virus reactivation, herpes zoster infection, pneumocystis pneumonia, etc), persistent hypogammaglobulinaemia, encephalopathy, severe neutropenia, fatal pulmonary fibrosis, ulcerative colitis, Crohn's disease and fulminant myocarditis etc. Adverse events will be graded according to the Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Qian Shen, Study Chair — Children's Hospital of Fudan University
Locations (3):
- China (3):
  - Children's hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai's Children's Medical Center, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to researchers with a clear research plan and hypothesis, with the appropriate team in place to undertake the work.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the article has been published with no end date
Access Criteria: Requests for access to data from the RTXFIRPedINS2 trial should be addressed to the corresponding author at hxu@shmu.edu.cn. The individual participant data collected during the trial (including the data dictionary) will be available, after de-identification. All proposals requesting data access will need to have a research plan and specify how the data will be used, and all proposals will need the approval of the trial coinvestigator team (or individual(s) subsequently delegated this responsibility) before data release

REFERENCES:
- [Result] Liu J, Shen Q, Xie L, Wang J, Li Y, Chen J, Fang X, Tang X, Qian B, Xu H. Protocol for an open-label, single-arm, multicentre clinical study to evaluate the efficacy and safety of rituximab in the first episode of paediatric idiopathic nephrotic syndrome. BMJ Open. 2022 Oct 12;12(10):e064216. doi: 10.1136/bmjopen-2022-064216. PMID 36223961